CLINICAL TRIAL: NCT06822998
Title: An Open-label, Single-arm, Non-randomized, Single-center, Dose-escalation Study to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of HF50 in Subjects With HER-2 Positive and HER-2 Low-expression Advanced Solid Tumors
Brief Title: HF50 in HER-2 Positive and Low-expression Advanced Solid Tumors
Acronym: HF50
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: HighField Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HF50-101
Record Dates: First submitted 2025-01-25; First posted 2025-02-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 - 1 mg (Experimental): Participants in this arm will receive HF50 via intravenous infusion once weekly for 3 weeks in a 3-week treatment cycle. The dose is 1 mg, with a lead-in dose on Cycle 1 Day 1 (C1D1) followed by the target dose on C1D8, C1D15, and C1D22.
  Interventions: Drug: HF50
- Dose Level 2 - 10 mg (Experimental): Participants in this arm will receive HF50 via intravenous infusion once weekly for 3 weeks in a 3-week treatment cycle. The dose is 10 mg, with a lead-in dose on C1D1 followed by the target dose on C1D8, C1D15, and C1D22.
  Interventions: Drug: HF50
- Dose Level 3 - 60 mg (Experimental): Participants in this arm will receive HF50 via intravenous infusion once weekly for 3 weeks in a 3-week treatment cycle. The dose is 60 mg, with a lead-in dose on C1D1 followed by the target dose on C1D8, C1D15, and C1D22.
  Interventions: Drug: HF50
- Dose Level 4 - 240 mg (Experimental): Participants in this arm will receive HF50 via intravenous infusion once weekly for 3 weeks in a 3-week treatment cycle. The dose is 240 mg, with a lead-in dose on C1D1 followed by the target dose on C1D8, C1D15, and C1D22.
  Interventions: Drug: HF50

INTERVENTIONS:
Drug: HF50 — HF50 is a liposomal T-cell engager with an unique design based on the lipid bilayer. It was also named a T cell Redirecting Antibody Fragment-anchored Liposomes (TRAFsome). The liposomal surface carries anti-CD3ε and anti-HER2 antibody-conjugated lipid molecules, enabling T-cell redirection and activation at HER2-positive or HER2-low tumor sites. In addition, the liposome internal space contains a TLR7/8 agonist Resiquimod (R848), which has been shown to help modulate the myeloid cells in the tumor micro-environement to complement the immune activation effects.

SUMMARY:
This is an open-label, single-arm, non-randomized, single-center, dose-escalation study designed to evaluate the safety and tolerability of HF50 in patients with HER-2 positive and HER-2 low-expression advanced solid tumors. The primary objectives are to assess the safety, tolerability, and determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of HF50. Secondary objectives include evaluating the pharmacokinetic (PK) profile and preliminary antitumor activity of HF50.

ELIGIBILITY:
Inclusion Criteria:

* Participants must voluntarily provide written informed consent (ICF) prior to any study-related procedures, and be capable of complying with all protocol requirements.
* Adult participants aged between 18 and 75 years (inclusive) at the time of ICF signing.
* Histologically or cytologically confirmed advanced HER-2 positive or HER-2 low-expression solid tumors that are unresectable, metastatic, or have relapsed after standard therapies, are intolerant to standard therapies (e.g., chemotherapy, targeted therapy), or lack effective treatment options.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 3 months.
* At least one measurable lesion as defined by RECIST version 1.1.
* Adequate organ and bone marrow function as demonstrated by the following laboratory parameters:Hematologic Function:Absolute neutrophil count (ANC) ≥1.5×10⁹/L、Lymphocyte count ≥1.0×10⁹/L、Platelet count ≥90×10⁹/L、Hemoglobin ≥9.0 g/dL (without transfusion or erythropoietin-stimulating agents within 14 days)； Coagulation Parameters:Activated partial thromboplastin time (aPTT) ≤1.5×ULN、 International normalized ratio (INR) ≤1.5. Hepatic Function:Total bilirubin (TBIL) ≤1.5×ULN、Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN for participants with liver metastases, and TBIL ≤3×ULN)； Renal Function:Creatinine clearance (CrCl) ≥50 mL/min (Cockcroft-Gault formula).
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and prior to the first dose. Male and female participants of childbearing potential must agree to use effective contraception during the study and for 6 months after the last dose.

Exclusion Criteria:

* History of active autoimmune disease or autoimmune disease considered unsuitable for study participation, with exceptions for localized skin conditions (e.g., eczema involving <10% of body surface area, vitiligo, psoriasis, alopecia) or childhood asthma resolved without treatment in adulthood.
* Current use of immunosuppressants or systemic corticosteroids (>10 mg/day prednisone or equivalent) within 4 weeks prior to the first dose, except for local steroid use.
* Receipt of systemic chemotherapy, radiotherapy, targeted therapy, or immunotherapy less than 2 weeks (or 4 weeks for nitrosourea or mitomycin C) or within 5 half-lives of the prior therapy before the first dose.
* Symptomatic brain metastases or leptomeningeal disease unless adequately treated (e.g., surgery or radiotherapy) with no evidence of progression for ≥28 days and off systemic steroids for ≥14 days prior to the first dose.
* Unresolved toxicities from prior therapies ≥Grade 2 (CTCAE v5.0) at baseline, except for toxicities deemed by the investigator to pose no safety risk (e.g., alopecia, stable hypothyroidism with hormone replacement).
* Significant cardiovascular or cerebrovascular conditions, including but not limited to:Thromboembolic events requiring therapeutic anticoagulation within 3 months prior to the first dose.NYHA Class III or IV heart failure.Acute coronary syndrome, congestive heart failure, aortic dissection, or stroke within 6 months prior to the first dose.Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg), unless controlled with antihypertensive medication.
* Active infection or unexplained fever >38.5°C within 1 week prior to the first dose (tumor-related fever may be eligible at the investigator's discretion).
* Known HIV infection, active hepatitis B virus (HBV) infection (HBV DNA >ULN), or active hepatitis C virus (HCV) infection (HCV RNA >ULN).
* Gastrointestinal symptoms or other conditions requiring intervention within 4 weeks prior to the first dose that would, in the investigator's judgment, impair study participation.
* Pregnant or breastfeeding women.
* Any other severe systemic disease, psychological condition, or significant clinical abnormality deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLT) | 28 days after the first dose (C1D1) for each dose cohort.
  The number of participants experiencing dose-limiting toxicities (DLTs) during the DLT evaluation period to determine the maximum tolerated dose (MTD).
Incidence of Adverse Events (AEs) | From first dose to 28 days after the last dose.
  The number and percentage of participants experiencing adverse events (AEs), graded according to NCI-CTCAE v5.0
Incidence of Serious Adverse Events (SAEs) | From first dose to 28 days after the last dose.
  The number and percentage of participants experiencing adverse events (AEs), graded according to NCI-CTCAE v5.0.
Recommended Phase II Dose (RP2D) of HF50 | At the end of dose escalation (assessed up to 1 year)
  RP2D will be determined based on safety, tolerability, and pharmacokinetics data collected during the dose escalation phase.
Incidence of Vital Sign Abnormalities | From first dose to the end of the study (assessed up to 1 year)
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline vital sign abnormality, including blood pressure, heart rate, respiratory rate, and body temperature. Grades are defined using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Laboratory Abnormalities | From first dose to the end of the study (assessed up to 1 year)
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including hematology (complete blood count), blood chemistry, urinalysis, coagulation function, and C-reactive protein (CRP). Grades are defined using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of Electrocardiogram (ECG) Abnormalities | From first dose to the end of the study (assessed up to 1 year)
  Number of participants who experienced an abnormal ECG finding post-baseline, including clinically significant changes in QT interval, PR interval, QRS duration, or other rhythm abnormalities as assessed by 12-lead ECG. Abnormalities will be graded according to National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of Echocardiography (ECHO) Abnormalities | From first dose to the end of the study (assessed up to 1 year)
  Number of participants who experienced an abnormal echocardiography finding post-baseline, including changes in left ventricular ejection fraction (LVEF), chamber size abnormalities, or valvular dysfunction. Abnormalities will be graded according to CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter - Cmax | Up to 9 weeks
  Maximum plasma concentration (Cmax) of HF50 will be assessed following single and multiple dosing.
Pharmacokinetic Parameter - Tmax | Up to 9 weeks
  Time to maximum plasma concentration (Tmax) of HF50 will be assessed following single and multiple dosing.
Pharmacokinetic Parameter - AUC (Area Under the Curve) | Up to 9 weeks
  AUC0-t and AUC0-inf will be evaluated to determine systemic exposure to HF50.
Pharmacokinetic Parameter - Half-life (t1/2) | Up to 9 weeks
  The terminal elimination half-life (t1/2) of HF50 will be calculated.
Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants achieving a complete response (CR) or partial response (PR) based on RECIST v1.1 criteria.
Duration of Response (DOR) | Up to 2 years
  Time from the first documented response (CR or PR) to disease progression or death.
Disease Control Rate (DCR) | Up to 2 years
  Proportion of participants achieving CR, PR, or stable disease (SD) based on RECIST v1.1.
Progression-Free Survival (PFS) | Up to 2 years
  Time from the first dose to disease progression or death.
Overall Survival (OS) | Up to 2 years
  Time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China